CLINICAL TRIAL: NCT03330665
Title: Meditation and Student Empathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BHS-1245
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Stress; Empathy
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No meditation
- Intervention (Experimental): Meditate using headspace app 3 times a week
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Meditation — Meditate 3 times a week using headspace app
  Other Names: MIndfullness
  Arms: Intervention

SUMMARY:
Physician empathy and reducing stress are major factors in attaining positive clinical outcomes for patients. Fostering empathy in medical students is particularly important as they are the future of the healthcare workforce and a trend of declining empathy during medical education may lead to decreased health care quality outcomes. Meditation may be an avenue to promote positive student attitudes including empathy, though very few studies have examined this idea through empirical research. Using validated measures, the Jefferson scale of empathy and the perceived stress scale, we seek to investigate whether use of a meditation app will be associated with higher levels of self-rated empathy and lower self-rated stress.

ELIGIBILITY:
Inclusion Criteria:

-Medical students from New York Institute of Technology

Exclusion Criteria:

-Not a medical student

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Perceived stress scale (PSS) | 6 months
  Perceived stress scale measures stress levels. 10 item scale where subjects are asked to indicate by circling how often they felt or thought a certain way on a scale of 1-4. Items are them added up- a higher score means higher stress.
Jefferson scale of empathy | 6 months
  Jefferson scale of Empathy measures empathy levels. 20 item scale where subjects are asked to indicate by circling how often they felt or thought a certain way about empathy related situations on a scale of 1-7. Items are them added up- a higher score means higher empathy.